CLINICAL TRIAL: NCT01091012
Title: Study About Effectiveness of the Vasodilator Test With Revatio, Made in Patients With Acute Pulmonary Hypertension, at Last Moderate and Secondary at Valve Disease(Corrected With a Normally Functioning Prosthesis).
Brief Title: Effectiveness of the Vasodilator Test With Revatio, Made in Patients With Acute Pulmonary Hypertension
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hospital Universitari Vall d'Hebron Research Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None
Other Study IDs: DOM-SIL-2009; 2009-012005-19 (EudraCT Number)
Record Dates: First submitted 2010-03-02; First posted 2010-03-23 (Estimated); Last update posted 2012-09-11 (Estimated); Status verified 2012-09

CONDITIONS: Pulmonary Hypertension
MeSH Terms: conditions — Hypertension, Pulmonary | interventions — Sildenafil Citrate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Sildenafil 20mg oral (Other)
  Interventions: Drug: Sildenafil 20mg oral vs Sildenafil 10mg intravenous
- Sildenafil 10mg intravenous (Other)
  Interventions: Drug: Sildenafil 20mg oral vs Sildenafil 10mg intravenous

INTERVENTIONS:
Drug: Sildenafil 20mg oral vs Sildenafil 10mg intravenous — 2 arms to comparation: Sildenafil 20mg oral vs intravenous Sildenafil 10mg
  Other Names: REVATIO oral vs REVATIO intravenous

SUMMARY:
The main objective is to validate the safety and efficacy of intravenous and oral sildenafil in the acute vasodilator test in patients with persistence of, at least, moderate pulmonary hypertension after valvular surgery successfully, with a correct left ventricular function and no valvular disease hemodynamically significant.

ELIGIBILITY:
Inclusion Criteria:

* Patients clinically stable, at least 1 year after the completion of successful valve surgery, with persistent pulmonary artery systolic pressure> 50 mmHg,
* normal left ventricular function and no significant valvular disease in 2 separate Doppler ultrasound studies at least 1 month.

Exclusion Criteria:

* Patients with other cardiac and noncardiac diseases will be excluded.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2011-09; Primary Completion 2012-12 (Estimated); Study Completion 2013-02 (Estimated)

PRIMARY OUTCOMES:
Effectiveness | one day per patient
  The main efficacy parameter is the effect on pulmonary vascular vasodilation quantified as decreased Pulmonary Vascular Resistance.

CONTACTS AND LOCATIONS:
Overall Officials: Enric Domingo, Promotor, Principal Investigator — Vall Hebron Hospital
Locations (1):
- Vall Hebron Hospital, Barcelona, Barcelona, Spain